CLINICAL TRIAL: NCT06231251
Title: Impact of Endoscopic Gastric Reduction of Ghrelin Receptors Rich Gastric Mucosa on Obesity and Metabolic Syndrome: a Randomized Controlled Trial
Brief Title: Endoscopic Gastric Reduction of Gastric Mucosa in Obesity
Acronym: ETO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Amr Shaaban Hanafy, professor of medicine and gastroenterology, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9352
Record Dates: First submitted 2022-06-30; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Obesity, Morbid; Endoscopy
MeSH Terms: conditions — Obesity, Morbid | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Intervention Model Description: endoscopic reduction of ghrelin rich gastric mucosa either with
  1. band ligation (group 1; n=16) and diet control
  2. argon plasma mediated reduction and diet control (group 2; n=16)
  3. control group exposed to low caloric diet and exercise (group 3; n=16).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Active Comparator): exposed to low caloric diet (15 calories/kilogram) and exercise
  Interventions: Other: upper gastrointestinal endoscopy
- endoscopic band ligation (Active Comparator): endoscopic reduction of ghrelin rich gastric mucosa with band ligation will be applied starting from the fundus till the mid body in 3-4 rows 1-2 cm apart for luminal reduction
  Interventions: Other: upper gastrointestinal endoscopy
- endoscopic argon plasma coagulation (Active Comparator): argon plasma mediated reduction of gastric mucosa rich in ghrelin receptors by appling argon to stomach mucosa from fundus to mid body
  Interventions: Other: upper gastrointestinal endoscopy

INTERVENTIONS:
Other: upper gastrointestinal endoscopy — reduction of ghrelin rich gastric mucosa with band ligation or argon plasma

SUMMARY:
In the stomach, the ghrelin-containing cells are more abundant in the fundus than in the pylorus originally termed X/A-like cells. These X/A-like cells account for approximately 20 % of the endocrine cell population in adult oxyntic glands.

Ghrelin enhances the secretion of growth hormone, the stimulation of appetite and food intake, the modulation of gastric acid secretion & motility and the endocrine and exocrine pancreatic secretions.

DETAILED DESCRIPTION:
Ghrelin is 28 amino acid peptide hormone, approximately 70 % of circulating ghrelin is secreted by the stomach, with most of the remainder originating in duodenum, jejunum, and ileum. Lower amount of secretion outside the gut, including hypothalamus (arcuate nucleus and paraventricular nucleus), pituitary, lung, adrenal cortex, kidney, bone, testis, placenta and pancreatic islet cells Ghrelin enhances the secretion of growth hormone, the stimulation of appetite and food intake, the modulation of gastric acid secretion & motility and the endocrine and exocrine pancreatic secretions. Synthetic ghrelin imitative was shown to increase fat deposition and appetite through an action at the level of the hypothalamus arcuate nucleus mainly the orexigenic neuropeptide Y (NPY) neurons.

Alterations of ghrelin play an important role in appetite fluctuation following meals. The secretion of ghrelin by the stomach depends largely on the nutritional state. Ghrelin levels show pre-prandial increases and postprandial decreases.

Low systemic ghrelin levels have been reported in untreated hyperthyroidism, in male hypogonadism, in the polycystic ovary syndrome, or after total gastrectomy [5, 6].

ELIGIBILITY:
Inclusion Criteria:

* body mass index more than 25
* diagnosis of diabetes mellitus.
* diagnosis of cardio-metabolic syndrome.
* fatty liver disease diagnosed by abdominal ultrasound.

Exclusion Criteria:

* use of drugs which induce insulin resistance, diabetes and hepatic steatosis.
* excess alcohol consumption.
* chronic gastritis, active peptic ulcer.
* malignancy.
* depression and severe psychological disorders
* inability to give informed consent.
* coagulopathy (INR more than 1.5, platelets less than 50000 per cmm).
* severe cardiopulmonary comorbidity.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-09-13 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with significant weight reduction | 6 month
  significant weight reduction of more than 10% of baseline body weight measured in kilograms

OTHER OUTCOMES:
Number of patients with improved insulin resistance | 6 months
  significant decrease in insulin resistance through assessing Homeostatic Model Assessment for Insulin Resistance, calculated by using the following formula: fasting glucose (mg/dL) X fasting insulin (µU/mL) / 405

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No